CLINICAL TRIAL: NCT00787137
Title: A Randomised, Double Blind, Placebo Controlled, Single Ascending Dose, Phase I Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of PG102 (Anti-CD40 Monoclonal Antibody) In Patients With Active Psoriatic Arthritis
Brief Title: Single Dose PG102 in Patients With Active Psoriatic Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: PanGenetics UK Limited (Industry)
Responsible Party: John Powell, PanGenetics UK Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PG102-01; 2007-001017-42 (EudraCT Number)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PG102 0.3 mg/kg (Experimental): Lowest dose PG102
  Interventions: Drug: PG102
- PG102 1 mg/kg (Experimental): Second dose PG102
  Interventions: Drug: PG102
- Placebo (phosphate-buffered saline) (Placebo Comparator): Control
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: PG102 — A single intravenous infusion
  Other Names: Anti-CD40 monoclonal antibody
  Arms: PG102 0.3 mg/kg; PG102 1 mg/kg
Drug: Placebo comparator — Phosphate-buffered saline
  Arms: Placebo (phosphate-buffered saline)

SUMMARY:
The primary objective is to evaluate the safety and tolerability of a single intravenous dose of PG102 in patients with psoriatic arthritis. The secondary objectives are to evaluate how PG102 moves around the body and to explore its effects on the disease.

ELIGIBILITY:
Inclusion Criteria:

* Arthritis that meets Classification of Psoriatic Arthritis (CASPAR) criteria
* Plaque psoriasis for at least 6 months prior to study enrollment

Exclusion Criteria:

* Clinically significant psoriasis flare
* Unstable doses of pain relief medication
* Treatment with systemic corticosteroids other than prednisone ≤ 10 mg/day or equivalent
* Treatment with any biologic therapy
* Treatment with immunosuppressive agents or disease modifying anti-rheumatic drugs (DMARDs) other than methotrexate
* Treatment with lithium, any anti-malarial, chlorambucil, cyclophosphamide or therapies for psoriasis other than low potency topical corticosteroids on intertriginous and groin areas, tar or salicylate preparations on the scalp, and emollients and moisturisers
* Family history of multiple thrombotic events or a personal history of any venous or arterial thrombotic event
* Clinically significant result for anti-cardiolipin, Activated protein C resistance test, Protein C, Free Protein S, Antithrombin III, Factor V Leiden, Prothrombin variant, Homocysteine, Lupus anticoagulant, Prothrombin time, Activated partial thromboplastin time, Fibrinogen, Thrombin time, Factors IX and XI
* Currently smoking ≥ 10 cigarettes per day or equivalent
* Active tuberculosis or other infection
* Current or previous malignancies
* Clinically significant abnormality on physical examination, laboratory testing, vital signs or 12-lead electrocardiogram

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nemanja Damjanov, MD PhD, Principal Investigator — Institute of Rheumatology, Belgrade, Serbia
Locations (1):
- Professor Nemanja Damjanov, Belgrade, Serbia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight study sites (rheumatology centres) in Serbia (3), Hungary (4) and the Russian Federation (1). The first patient's first visit was on December 2, 2008 and the last visit for the last patient was on April 21, 2010.
Pre-assignment Details: The first three patients in each cohort were dosed sequentially and could not be taking methotrexate. Subsequent patients in each cohort could be dosed simultaneously and could be taking methotrexate. There was a pause between dosing the last patient in the first cohort and the first patient in the second cohort.
Groups:
- Placebo: Control, phosphate-buffered saline
Period: Overall Study
Arm/Group | PG102 0.3 mg/kg | PG102 1 mg/kg | Placebo
Started | 6 | 6 | 5
Completed | 6 | 6 | 4
Not Completed | 0 | 0 | 1
Not completed — Study Termination | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PG102 0.3 mg/kg | PG102 1 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 5 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 5 | 17
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Full Range); unit: years] | 43.3 (9.77) [32 to 54] | 43.8 (10.85) [27 to 59] | 45.2 (13.20) [31 to 58] | 44.0 [27 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 5 | 6 | 4 | 15
Region of Enrollment [Number; unit: Participants]
  Serbia | 2 | 5 | 2 | 9
  Hungary | 4 | 1 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Reported Adverse Events
Description: This was an exploratory study and all safety endpoints were considered.
Time Frame: Three months
Population: All adverse events reported for all patients dosed were evaluated
Measure: Number; unit: Number of adverse events
Arm/Group | PG102 0.3 mg/kg | PG102 1 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Number of adverse events | 3 | 6 | 13

2. Primary Outcome: The Percentage of Participants With Adverse Events
Time Frame: Three months
Population: All patients dosed were evaluated
Measure: Number; unit: Percentage of Participants
Arm/Group | PG102 0.3 mg/kg | PG102 1 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Percentage of Participants | 50 | 67 | 40

3. Primary Outcome: The Number of Episodes of Change in Vital Signs
Description: Clinically significant episodes of change in blood pressure, heart rate, temperature or respiration rate on the day before dosing and 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours and 4, 7, 14, 21, 28, 56 & 84 days after dosing. The investigator evaluated clinical significance primarily by blinded comparison with the respective screening value.
Time Frame: Three months
Measure: Number; unit: Number of episodes of change
Arm/Group | PG102 0.3 mg/kg | PG102 1 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Number of episodes of change | 0 | 0 | 1

4. Primary Outcome: The Number of Episodes of Change in Electrocardiogram
Description: Episodes of clinically significant change in 12-lead electrocardiogram predose,1 & 4 hours and 1 & 84 days postdose. The investigator evaluated clinical significance primarily by blinded comparison with the screening electrocardiogram.
Time Frame: Three months
Measure: Number; unit: Number of episodes of change
Arm/Group | PG102 0.3 mg/kg | PG102 1 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Number of episodes of change | 0 | 0 | 0

5. Primary Outcome: The Number of Episodes of Change From Screening in Laboratory Assessments
Description: Red cell count, haemoglobin, haematocrit, total and differential white cell counts, platelet count, mean corpuscular volume, mean corpuscular haemoglobin, mean corpuscular haemoglobin concentration, reticulocytes; urea, creatinine, urate, bilirubin, sodium, potassium, calcium, phosphate, chloride, bicarbonate, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, gammaglutamyl transferase, creatine phosphokinase, albumin, protein; urine pH, protein, glucose, ketones, bilirubin, blood, urobilinogen, nitrite, leucocytes, specific gravity.
Time Frame: Three months
Measure: Number; unit: Number of episodes of change
Arm/Group | PG102 0.3 mg/kg | PG102 1 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Number of episodes of change | 4 | 7 | 3

ADVERSE EVENTS:
Arm/Group | PG102 0.3 mg/kg | PG102 1 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG102 0.3 mg/kg (N=6) | PG102 1 mg/kg (N=6) | Placebo (N=5)
Transaminases increased/hepatic enzymes increased (Investigations) | 1 (1) | 4 (4) | 0 (0) — The term for transaminases increased and hepatic enzymes increased have been grouped together because the events were comparable in ALT/AST ratio, involvement or lack of involvement of other analytes and in time of onset.
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Leucocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Termination prior to accrual of planned numbers of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An investigator shall not publish any data (poster, abstract, paper etc) without having consulted with the Sponsor in advance.